CLINICAL TRIAL: NCT06808659
Title: Comparative Effects of Neural Mobilization of Sciatic Nerve Versus Stretching Among Patients With Piriformis Syndrome
Brief Title: Effects of Neural Mobilization and Stretching in Piriformis Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Rabia Khan, Assistant Professor, Bahria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IERC/IIRS-IU-KC/18/005
Record Dates: First submitted 2024-11-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Piriformis Syndrome
Keywords: Physiotherapy; Piriformis Stretching; Visual Analog Scale (VAS); Pain Management; FAIR Test; Range of Motion
MeSH Terms: conditions — Piriformis Muscle Syndrome; Agnosia

STUDY DESIGN:
Intervention Model Description: In a study involving 40 patients diagnosed with sciatica, researchers aimed to investigate whether neural mobilization of the sciatic nerve or stretching of the piriformis muscle was more effective in treating piriformis syndrome. The patients were divided into two groups, each containing 20 individuals. Group A underwent neural mobilization therapy, while Group B performed piriformis muscle stretches, with both groups receiving treatment three times a week for two weeks. Assessments, including Visual Analog Scale (VAS) for pain, hip range of motion (ROM) in flexion, abduction, and external rotation, as well as the FAIR test, were conducted before and after the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A / Sciatic Nerve Mobilization (Experimental): Sciatic Nerve Mobilization was given to group A participants.
  Interventions: Other: Neural Mobilization
- Group B / Piriformis Muscle Stretching (Experimental): Piriformis Muscles was stretched in group B participants.
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Neural Mobilization — A total of 20 patients were selected in Group A received neural mobilization of sciatic nerves treatment for 3 days a week for 2 weeks
  Other Names: Sciatic Nerve Mobilization
  Arms: Group A / Sciatic Nerve Mobilization
Other: Stretching — A total of 20 patients were selected in Group B received stretching of piriformis muscle treatment for 3 days a week for 2 weeks
  Other Names: Piriformis Stretching
  Arms: Group B / Piriformis Muscle Stretching

SUMMARY:
This study compares the effects of piriformis stretching and neural mobilization of the sciatic nerve in individuals with piriformis syndrome, a condition that is frequently characterized by hip and buttock pain and discomfort brought on by the piriformis muscle compressing the sciatic nerve.

DETAILED DESCRIPTION:
In a study involving 40 patients diagnosed with sciatica, researchers aimed to investigate whether neural mobilization of the sciatic nerve or stretching of the piriformis muscle was more effective in treating piriformis syndrome. The patients were divided into two groups, each containing 20 individuals. Group A underwent neural mobilization therapy, while Group B performed piriformis muscle stretches, with both groups receiving treatment three times a week for two weeks. Assessments, including Visual Analog Scale (VAS) for pain, hip range of motion (ROM) in flexion, abduction, and external rotation, as well as the FAIR test, were conducted before and after the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Positive lasegue sign
* Positive piriformis sign
* Tenderness at sciatic notch (over piriformis muscle).

Exclusion Criteria:

* • Prior surgery of lumbar spine (laminectomy)

  * Unrecognized pelvic fracture
  * Known case of renal stones
  * Disc herniation in lumbar spine
  * Myositis ossificans of piriformis muscle.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Pain Reduction | 2 weeks
  Two different interventions were applied in groups after which pain was recorded before and after through visual analogue scale. Highest score means high level of pain and lower score refers to low pain. Maximum score 9 was reported pre study and minmum score 2 was reported after study by both groups on average.
Increase Range of Motion | 2 weeks
  Through neural mobilization and piriformis stretching renage of motion was assessed through inclino meter before and after study

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Khan, Masters of Science, Principal Investigator
Locations (1):
- Isra Institute of Rehabilitation Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Confidentiality

REFERENCES:
- [Background] Othman IK, Raj NB, Siew Kuan C, Sidek S, Wong LS, Djearamane S, Loganathan A, Selvaraj S. Association of Piriformis Thickness, Hip Muscle Strength, and Low Back Pain Patients with and without Piriformis Syndrome in Malaysia. Life (Basel). 2023 May 18;13(5):1208. doi: 10.3390/life13051208. PMID 37240853
- [Background] Hu YE, Ho GWK, Tortland PD. Deep Gluteal Syndrome: A Pain in the Buttock. Curr Sports Med Rep. 2021 Jun 1;20(6):279-285. doi: 10.1249/JSR.0000000000000848. PMID 34099604
- [Background] Danazumi MS, Yakasai AM, Ibrahim AA, Shehu UT, Ibrahim SU. Effect of integrated neuromuscular inhibition technique compared with positional release technique in the management of piriformis syndrome. J Osteopath Med. 2021 May 31;121(8):693-703. doi: 10.1515/jom-2020-0327. PMID 34049428
- [Background] Burke CJ, Walter WR, Adler RS. Targeted Ultrasound-Guided Perineural Hydrodissection of the Sciatic Nerve for the Treatment of Piriformis Syndrome. Ultrasound Q. 2019 Jun;35(2):125-129. doi: 10.1097/RUQ.0000000000000360. PMID 29727344
- [Background] Shahzad M, Rafique N, Shakil-Ur-Rehman S, Ali Hussain S. Effects of ELDOA and post-facilitation stretching technique on pain and functional performance in patients with piriformis syndrome: A randomized controlled trial. J Back Musculoskelet Rehabil. 2020;33(6):983-988. doi: 10.3233/BMR-181290. PMID 32894238
- [Background] Ahmad Siraj S, Dadgal R. Physiotherapy for Piriformis Syndrome Using Sciatic Nerve Mobilization and Piriformis Release. Cureus. 2022 Dec 26;14(12):e32952. doi: 10.7759/cureus.32952. eCollection 2022 Dec. PMID 36712711
- [Result] Ankar P, Ratnani GR, Ramteke SU, Jaiswal PR. Effect of Neuromuscular Training and Neurodynamic Solutions for Asymptomatic Prolapsed Intervertebral Disc and Coexisting Piriformis Syndrome in a 19-Year-Old: A Comprehensive Case Report. Cureus. 2024 Jan 27;16(1):e53050. doi: 10.7759/cureus.53050. eCollection 2024 Jan. PMID 38410291
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/?term=effect%20of%20piriformis%20syndrome%20on%20pain%20&filter=dates.2018%2F4%2F10-2023%2F12%2F30&page=3